CLINICAL TRIAL: NCT05061329
Title: The Importance of the Nasal Microbiome in Transmission and Disease
Brief Title: The Nasal Microbiome and Its Importance in Disease
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: NasalMicrobiomeTO,LD,KF
Record Dates: First submitted 2021-09-21; First posted 2021-09-29 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Chronic Rhinosinusitis (Diagnosis); COVID-19; Anosmia
MeSH Terms: conditions — Disease; COVID-19; Anosmia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Microbiome swabs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 60 Normal individuals: Normal sense of smell and absence of sino-nasal disease, upper airway allergies, and no intranasal medication
- 60 Non-COVID-19 positive patients: with olfactory dysfunction
- 15 COVID-19 positive patients: In the acute phase
- 60 long COVID-19 patients: with olfactory dysfunction persisting for more than 12 weeks
- 60 patients with chronic rhinosinuitis: initiating intranasal glucocorticoids
- 15 patients with chronic rhinosinuitis: initiating biological treatment with either dupilumab or mepolizumab

SUMMARY:
Methods: all studies are case control studies on six different groups: normal individuals, non-COVID-19 patients with olfactory dysfunction, COVID-19 positive patients, previous COVID-19 positive patients with prolonged olfactory dysfunction, patients with chronic rhinosinusitis with and without nasal polyps, and patients with CRS initiating intranasal glucocorticoids.. The patients will be included from the ear-, nose, and throat department and the University Clinic for Flavour, Balance, and Sleep Regional Hospital Gødstrup, as well as Flavour Institute, Department of Clinical Medicine, Aarhus University (AU), and the long COVID-19 clinics in Aarhus and Gødstrup.

Microbiome samples will be swabs from the nasal cavity and oral pharynx will be collected and analysed using next-generation sequencing targeting 16S and 18S ribosomal RNA at the Department of Bacteria, Parasite & Fungi at Staten Serum Institute (SSI), Copenhagen, Denmark. Characterization of the microbiome is performed by 16S/18S amplicon-based metagenomics, and data are analyzed by various bio-informatic tools for determination/visualization of alpha/beta diversity as well as principal coordinates analysis (PCoA). Immunological factors will be collected by means of six swabs: in the nasal cavity and used for either flowcytometry or enzyme-linked immunosorbent assay (ELISA).

For comparison, truecut biopsies of the nasal mucosa are collected from a subgroup of patients undergoing surgery in general anaesthesia.

Due to the novelty of the current study, little relevant information from previous literature can be used for power calculation. However, with an alpha of 5% and a power of 80%, the population size for each group should be 42 participants, assuming the occurrence of bacteria differs with 30% between populations. Taking 20% drop out into account, the investigators aim to include 60 patients in each group.

Perspectives:

The perspectives of this study is to begin bridging the gap between gut and upper airway microbiome and immunology research. Looking at the explosion of interest in the gut, and in personalized medicine in general, the investigators likewise foresee a huge potential for both general and individual prevention and treatments starting with a deeper understanding of the nasal microbiome and immunology. Examples beyond the scope of this study could be microbiome transplants for chronic sufferers of diseases such as chronic rhinosinusitis, allergies or asthma, or in selecting which patients could reap the benefits of the expensive biological treatments emerging on the market.

DETAILED DESCRIPTION:
Hypotheses

The following null hypotheses are suggested:

1. The nasal microbiome in patients with olfactory dysfunction does not differ from healthy individuals with normal olfaction
2. Seasonal fluctuations in the nasal microbiome do not occur
3. The immunologic landscape of the nasal mucosa does not correlate with specific microbi-omes
4. Neither intranasal glucocorticoids nor dupilumab and mepolizumab affect the nasal mi-crobiome and local immune factors in patients with CRSwNP Materials and methods Design: Case-control study and longitudinal cohort study.

Populations:

1. 60 healthy controls: Normal sense of smell and absence of sino-nasal disease, upper air-way allergies, and no intranasal medication
2. 60 non-COVID-19 patients with olfactory dysfunction
3. 15 COVID-19 positive patients in the acute phase
4. 60 long COVID-19 patients with olfactory dysfunction persisting for more than 12 weeks
5. 60 patients with CRS initiating intranasal glucocorticoids
6. 15 patients with CRS initiating biological treatment

Inclusion criteria

- Older than 18 years

Exclusion criteria

* For the biopsy groups, active anticoagulation treatment
* Diseases of the coagulant system
* Antibiotics in the last three months
* Other immunomodulating drugs in the last three months
* Autoimmune disease or immunodeficiency

Recruitment: Population 1, 5, and 6 are recruited among patients undergoing sino-nasal surgery at the ear-nose-throat department, Regional Hospital Gødstrup, Denmark. Populations 2 and 4 are enrolled from the Flavour Institute, Department of Clinical Medicine, Aarhus University, Denmark, and University Clinic for Flavour, Balance, and Sleep, Gødstrup Regional Hospital, Denmark. Popu-lation 3 is recruited at the long COVID-19 clinics at Aarhus University Hospital and at Gødstrup Regional Hospital. Population 1 will be supplied with staff members and university students.

Clinical examinations, measurements and information: For all participants, information is ob-tained on medical history, medicine use, objective ear, nose, and throat examination including endoscopy of upper airways, Sino-Nasal Outcome Test-22[9], Major Depression Inventory[10,11], Mini Mental Status[12], Sniffin' Sticks[13], and taste screening.

Microbiome samples: Swabs from the nasal cavity and oral pharynx will be collected for microbi-ome analysis using next-generation sequencing targeting 16S and 18S ribosomal RNA. Characteri-zation of the microbiome is performed by 16S/18S amplicon-based metagenomics, and data are analyzed by various bioinformatic tools for determination/visualization of alpha/beta diversity as well as principal coordinates analysis (PCoA).

Intranasal immune factors: Nasal biopsies (3x3x3 mm) will be characterized histologically and analysed using spatial transcriptomics on the Vision 10X Genomics platform. Nasal secretion is collected by means of six swabs and used to characterize the cytokine profile. A broad Luminex-based panel encompassing 45 cytokines and chemokines will be employed (Invitrogen, Cyto-kine/Chemokine/Growth Factor Convenience 45-Plex Human ProcartaPlex™ Panel 1), and samples will be run in duplicate. The panel includes cytokines known to play a role in CRS, and which are targeted by biologic treatment, such as IL-4, IL-13, and IL-5.

Data on nasal steroid use: Patients starting intranasal glucocorticoids will be included upon com-mencement of treatment and follow up will be after 24 weeks.

Statistics: With an alpha of 5% and a power of 80%, the population size for each group should be 42 participants, assuming the occurrence of bacteria differs with 30% between populations. Tak-ing 20% drop out into account, the investigators aim to include 60 patients in group 1-4. The studies involving group 5 and 6 are explorative and hypothesis-generating, and power calculations have not been performed. Furthermore, only few patients fulfil the criteria for biological treatment; hence the investigators intend to include all patients initiating biological treatment within 12-18 months.

Feasibility: The project is a collaboration between the applicant; professor, senior consultant, DMSc, Therese Ovesen, Flavour Institute, Aarhus University & The Flavour Clinic, Gødstrup Re-gional Hospital; and senior consultant, DMSc, Kurt Fuursted, Statens Serum Institute (SSI). The Flavour Institute, receives patients from all over Denmark, and since 2015 almost 3000 patients have consulted the unit, and more than 50 research studies of olfactory dysfunction have been published from the Flavour Clinic and Institute. Since 2016, routine clinical microbiome diagnos-tics, 16S/18S amplicon-based metagenomics, has been conducted at SSI, and both clinical and bioinformatic expertise will be provided in this field by SSI. The project further leverages a collab-oration with the CellX initiative housed at MOMA, which is a national initiative providing expertise and infrastructure for single-cell omics. Overall, the investigators vouch for both the required number of pa-tients, and a solid and extensive experience with all test methods, equipment, and the necessary infrastructure.

The regulatory requirements for Study 1 and 2 are in place and patient enrollment as well as microbiome sample collection has already begun.

Ethics: None of the smell or taste tests, nor sampling of microbiome and immune factors causes danger, discomfort or pain. GDPR is complied with in all studies and data is stored on computers following legal requirements. The study fulfills the Helsinki declaration and is approved by the local ethic committee (reg.nr. 1-10-72-213-21). Regarding nasal biopsies, this is routine work up in ENT outpatient clinics. The biopsy is taken from middle turbinate in local anesthesia and measures 3x3x3 mm. An additional application for permission to obtain the biopsies will be send to the local ethical committee. The risk of bleeding is very low as patients with hematological diseases and patients in anticoagulant therapy are excluded.

The microbiome will be evaluated using swabs from the nasal cavity and analysed using next-generation sequencing targeting 16S and 18S ribosomal RNA at the Department of Bacteria, Parasite & Fungi at Staten Serum Institute, Copenhagen, Denmark.

Nasal biopsies (3x3x3 mm) will be characterized histologically and analysed using spatial tran-scriptomics on the Vision 10X Genomics platform. Nasal secretion is collected by means of six swabs and used to characterize the cytokine profile.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Does not wish to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Normal individuals: no sino-nasal disease - no upper airway allergies - no intra nasal medication - normal sense of smell
  2. Patients with smell loss
  3. COVID-19 positive patients
  4. Previous COVID-19 positive patients with prolonged olfactory dysfunction
  5. Patients with chronic rhinosinusitis with and without nasal polyps
  Recruitment: population 1, 5, and 6 are recruited among patients undergoing surgery at the ENT department, Regional Hospital West Jutland, Denmark. Populations 2 and 4 are enrolled from the Flavour Clinic, ENT department, Regional Hospital Denmark. Population 3 is recruited at the COVID-19 clinics in Aarhus and Herning. Population 1 will be supplied with staff members and university students.
Sampling Method: Non-Probability Sample
Enrollment: 619 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome difference | 6 months
  Difference in microbiome between the defined groups

SECONDARY OUTCOMES:
Effect of nasal glucocorticoids on nasal microbiome | 6 months
Correlation between TDI score and nasal microbiome | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Marie Aalkjær Danielsen, Principal Investigator — student
Locations (1):
- Ear, Nose and Throat Department, HEV, Holstebro, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided